CLINICAL TRIAL: NCT01954368
Title: Acute Severe Traumatic Pain in the ED : Can we Improve Time to Pain-relief With a Single Dose of Intranasal Sufentanil Given at Triage ? A Randomized Double-blinded Placebo Controlled Study (InSPEED Study)
Brief Title: Intranasal Sufentanil Pain-management at Entrance of Emergency Department : Influence on Pain-relief Delay
Acronym: InSPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-AOI-10; 2013-003308-38 (EudraCT Number)
Record Dates: First submitted 2013-09-20; First posted 2013-10-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Single Traumatic Limb Injury With Severe Pain (Score > 5/10 on Numerical Pain Scale)
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intranasal placebo (Placebo Comparator): Patients receiving intranasal placebo at ED admission
  Interventions: Drug: Placebo
- Intranasal sufentanil (Experimental): Patients receiving intranasal sufentanil at ED admission
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Placebo — As soon as possible from ED admission, using a study drug volume schedule, triage nurse will administer to the patient a planned weight-based volume of intranasal placebo (normal saline solution).
  Half of the dose will be administrated in each nostril. The patient will then rapidly be brought to emergency room and after his pain being reassessed, appropriate treatment (following current recommendations) will be given by the ED nurse.
  Arms: Intranasal placebo
Drug: Sufentanil — As soon as possible from ED admission, using a study drug volume schedule, triage nurse will administer to the patient a weight-based volume (corresponding to 0,4 mcg/kg) of intranasal sufentanil.
  Half of the dose will be administrated in each nostril. The patient will then rapidly be brought to emergency room and after his pain being reassessed, appropriate treatment (following current recommendations) will be given by the ED nurse.
  Arms: Intranasal sufentanil

SUMMARY:
Non-invasive and simple, intranasal (IN) route of administration seems promising for pain management in the Emergency Department (ED), especially when used precociously by triage nurse to rapidly deliver the first opioid dose to severely painful patients.

This randomized double-blind placebo-controlled study will focus on severe traumatic pain experienced by adults admitted in our ED.

We hypothesized that, in addition to traditional morphine titration, a single dose of IN sufentanil given at triage would significantly increase the proportion of patients relieved 30 minutes after their ED admission.

Time to discharge, proportion of side effects and satisfaction rates will also be recorded.

DETAILED DESCRIPTION:
Time to pain-relief can vary widely in the Emergency Department (ED), depending on various factors such as ED overcrowding or inadequate training in pain management.

As intravenous (IV) opioid administration is world-wide recommended for severe pain treatment, delays from triage to room admission and to first IV injection directly influence this time to pain-relief. Moreover, it is proven that an incorrect adherence to morphine titration protocol can participate in ED oligoanalgesia.

Although ED experience in intranasal (IN) opioid administration is still lacking, this simple and non-invasive way of treating pain seems safe and promising. Opioid pharmacokinetic by IN route indeed is interesting for ED practitioners : while assuring a timely analgesia, the lower Cmax and delayed Tmax by IN route can theoretically limit the risk of respiratory depression, in comparison with IV route.

We propose a randomized double-blind placebo-controlled study on a convenience sample of adult patients admitted in our ED (annual census of 80000 attendances) for an isolated limb injury, and experiencing a severe pain (score > 5/10 on numerical pain scale).

For primary outcome, we will compare the proportion of patients relieved (score < 4/10) 30 minutes after admission, depending on the administration (or not) of a single intranasal dose of sufentanil (0,4 mcg/kg) given by the triage nurse.

Other secondary outcomes will include : evolution of pain scores in the first hour of admission and during entire ED stay, proportions of opioid-induced side-effects, proportions of patients receiving morphine and doses of morphine administrated, times for discharge, patient and staff satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* Single traumatic limb injury.
* Severe pain (score > 5/10 on numerical pain scale)
* Age ≥ 18 years and < 75 years

Exclusion Criteria:

* Abdominal, thoracic, vertebral or cranial injury associated
* Hemodynamic instability (systolic blood pressure < 100 mmHg and/or blood pulse > 110 / min)
* Oxygen saturation < 96% on room air
* Chronic respiratory, renal or cardiac failure
* Impaired mental status (Glasgow Coma Scale < 15)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pain relief assessment | 30 minutes after ED admission
  Proportion of patients pain-relieved (score < 4/10 on numerical pain scale) at T30 (30 minutes after their admission)

SECONDARY OUTCOMES:
opioids-related side-effects | 2h after last opioid injection.
  Proportions of opioids-related side-effects.
Pain assessment | 30 minutes after ED admission
  Proportions of patients having a score on numerical pain scale < 6/10 at room admission.
time to pain relief treatment | 30 minutes after ED admission
  Delay from ED admission to first opioid injection (IV morphine or IN sufentanil).
Delay from first opioid injection to pain-relief | 30 minutes
  Delay from first opioid injection (IV morphine or IN sufentanil) to pain-relief.
Patient satisfaction | at discharge
  Patient satisfaction score at discharge (an average time of 12h) (on a " zero-to-10 " scale)
ED length of stay | 8 h after ED admission
  ED length of stay.
Nurse satisfaction | at discharge
  Nurse satisfaction score at discharge (an average time of 12h)(on a " zero-to-10 " scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Department, Nice, France